CLINICAL TRIAL: NCT00581763
Title: Long-Term Outcome of Children and Adolescents With Anti-Phospholipid Antibodies
Acronym: APL
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: H8994-19045
Record Dates: First submitted 2007-12-19; First posted 2007-12-28 (Estimated); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Lupus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Observation: Those with a condition

SUMMARY:
This is a study about why some people have certain types of proteins in their blood, called anti-phospholipid antibodies. The presence of these antibodies and associated complications (e.g. blood clots) are known to change over time. The purpose of this study is to evaluate these changes and improve our ability to determine the long-term outcome of affected individuals.

DETAILED DESCRIPTION:
Aim:

1. Determine the incidence, and time frame, for aquiring aPL in a cohort of aPL-negative pediatric SLE subjects.
2. Determine the incidence, and time frame, for developing a first APS-associated complication among SLE subjects with detectable aPL.
3. Determine the incidence, and time frame, for developing a second APS-associated event among subjects with a history of an APS-associated event.
4. Determine the incidence, and time frame, for developing SLE among subjects with a history of an APS-associated event in the absence of SLE.
5. Identify laboratory and clinical predictors for the events described in aims 1-4.Research Design and Methods:

This is a prospective cohort study to determine the risk of developing aPL or APS-related symptoms in a young group of SLE and APS subjects. Patients will be followed over a ten year period and will undergo annual serologic and clinical evaluations to identify disease progression.

ELIGIBILITY:
Inclusion Criteria:

Age: Less than 21 years at baseline exam

* Diagnosis: patients must meet criteria for one of five diagnostic categories based on classification according to three parameters; aPL positivity, APS criteria, and SLE criteria.

The five diagnostic categories are:

* SLE with no aPL
* SLE with aPL, but without manifestations of APS
* SLE-like APS
* SLE with APS
* Primary APS.

Exclusion Criteria:

* none

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Young group of SLE and APS subjects
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2001-05; Primary Completion 2019-12-20 (Actual); Study Completion 2019-12-20 (Actual)

PRIMARY OUTCOMES:
thrombosis | Ten years
  blood clot

SECONDARY OUTCOMES:
lupus | 10 years
  systemic lupus erythematosus

CONTACTS AND LOCATIONS:
Overall Officials: Emily von Scheven, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States